CLINICAL TRIAL: NCT02765074
Title: Filling Bone Erosions: a Longitudinal Multicentric HR-pQCT Study of 12 Months Subcutaneous Tocilizumab in Rheumatoid Arthritis Phase IV Prospective Multicentrique Study
Brief Title: Filling Bone Erosions: a Longitudinal Multicentric HR-pQCT Study of Subcutaneous Tocilizumab in Rheumatoid Arthritis
Acronym: REPAIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Collaborators: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHRO 2014-03
Record Dates: First submitted 2016-04-19; First posted 2016-05-06 (Estimated); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis
Keywords: subcutaneous tocilizumab; High Resolution peripheral QCT (HR-pQCT); bone erosion; bone microarchitecture; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Roactemra (Experimental): subcutaneous tocilizumab
  Interventions: Drug: subcutaneous tocilizumab

INTERVENTIONS:
Drug: subcutaneous tocilizumab — 162 mg subcutaneous, once a week during 12 months
  Other Names: Roactemra

SUMMARY:
Rheumatoid arthritis (RA) is a chronic inflammatory disease mediated by the production of several cytokines, which leads to the destruction of bone and cartilage tissue in multiple joints and to bone loss. Conventional radiographs (CR) are considered as the gold standard for diagnosis and follow up of joint changes in RA. But this method has low sensitivity to detect early erosive changes and is unable to evaluate periarticular bone loss.

High Resolution peripheral QCT (HRpQCT) enables the detection of erosions less than 0.5 mm in width or depth at metacarpo-phalangeal (MCP) joints. Using 3-D high resolution analysis of cortical bone erosions, this one is also able to evaluate the volumes of erosion and the evolution under treatments IL6 (6- interleukin) plays a major role in inflammatory process and bone damages related to RA. Tocilizumab (TCZ) is a humanized anti-IL-6R monoclonal antibody, developed and investigated in several clinical trials in RA. This biotherapy, in association with methotrexate (MTX) or given in monotherapy, is efficient in RA with inadequate response to MTX or anti-TNF b (tumor necrosis factor). TCZ reduces dramatically systemic inflammation, structural progression and improves clinical symptoms and quality of life.

Tocilizumab may help reducing bone erosions, periarticular osteopenia and systemic bone loss.

ELIGIBILITY:
Inclusion Criteria:

* Active RA, < 10 years disease duration, diagnosed according to the ACR-EULAR 2010 classification criteria
* DAS 28 superior or equal to 3.2 despite DMARD or biological treatment (other than tocilizumab)
* Superior or equal to one joint erosion at the right or left MCP 2, 3 on X-rays
* Oral corticosteroid ≤ 10 mg/day prednisone or equivalent stable for at least one month
* RA patients eligible to subcutaneous Tocilizumab monotherapy

Exclusion Criteria:

* Treatment with zoledronic acid or denosumab (less than one year)

  * Intra-articular injection of corticosteroids at the MCP in the previous three months
  * Tocilizumab contra-indications in accordance with SPC (Summary of Product Characteristics) :Hypersensitivity to the active substance or to any of the excipients Active, severe infections including active tuberculosis Diverticulitis Active hepatic disease and hepatic Impairment including viral hepatitis Elevated Alanine Aminotransferase or Aspartate Aminotransferase >5×ULN Absolute neutrophil count < 0.5 × 10 exp 9 /L Platelet count < 50×10 exp 3 /μL,

General:

* Absence of informed consent
* Prior or planned joint surgery of the hands which might impact the interpretation of imaging assessments.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Bone erosion change after 12 months of subcutaneous tocilizumab | baseline and 12 months
  changes of width measured by HRpQCT.
Bone erosion change after 12 months of subcutaneous tocilizumab | baseline and 12 months
  changes of depth measured by HRpQCT.
Bone erosion change after 12 months of subcutaneous tocilizumab | baseline and 12 months
  changes of volume measured by HRpQCT.

SECONDARY OUTCOMES:
Associated factors with erosion changes assessed by HRqQCT | baseline, 3 months, 12 months
  Number of participants with associated factors with erosion changes by HRpQCT (Associated therapeutic, clinical and biological response )ultrasound ...)
Effect of 12 months of tocilizumab on bone density in the PR | baseline, 12 months
  Changes of Bone mineral density by DXA at the lumbar spine and proximal femur
Effect of Tocilizumab on synovitis/tenosynovitis assessed by US and agreement with disease activity scores | Predictors baseline, 1 and 3 months of clinical remission and / or ultrasound at 6 and 12 months
  Correlation Between clinical activity measured by various indices (Disease Activity Score 28, Clinical Disease Activity Iindex , Simplify Disease Activity Index , American College of Rheumatology - European League against Rheumatism: ACR EULAR) and ultrasound data.
Effect of 12 months of tocilizumab on bone microarchitecture in the PR | baseline, 12 months
  changes of bone microarchitecture by tibia HRpQCT

CONTACTS AND LOCATIONS:
Overall Officials: SALLIOT Carine, MD, Study Director — CHR ORLEANS; LESPESSAILLES Eric, MD, PhD, Principal Investigator — CHR ORLEANS; CANTAGREL Alain, MD, PhD, Principal Investigator — University Hospital, Toulouse; CHAPURLAT Roland, MD, PhD, Principal Investigator — Hospices Civils de Lyon; MAROTTE Hubert, MD, PhD, Principal Investigator — HOPITAL NORD SAINT ETIENNE
Locations (4):
- France (4):
  - Hopital Edouard HERIOT, Lyon
  - CHR d'ORLEANS, Orléans
  - Hopital Nord CHU de SAint ETIENNE, Saint-Etienne
  - Chu Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boutroy S, Bouxsein ML, Munoz F, Delmas PD. In vivo assessment of trabecular bone microarchitecture by high-resolution peripheral quantitative computed tomography. J Clin Endocrinol Metab. 2005 Dec;90(12):6508-15. doi: 10.1210/jc.2005-1258. Epub 2005 Sep 27. PMID 16189253
- [Background] Stach CM, Bauerle M, Englbrecht M, Kronke G, Engelke K, Manger B, Schett G. Periarticular bone structure in rheumatoid arthritis patients and healthy individuals assessed by high-resolution computed tomography. Arthritis Rheum. 2010 Feb;62(2):330-9. doi: 10.1002/art.27252. PMID 20112404
- [Background] Fouque-Aubert A, Boutroy S, Marotte H, Vilayphiou N, Bacchetta J, Miossec P, Delmas PD, Chapurlat RD. Assessment of hand bone loss in rheumatoid arthritis by high-resolution peripheral quantitative CT. Ann Rheum Dis. 2010 Sep;69(9):1671-6. doi: 10.1136/ard.2009.114512. Epub 2010 Jun 4. PMID 20525847
- [Background] Ellouz R, Chapurlat R, van Rietbergen B, Christen P, Pialat JB, Boutroy S. Challenges in longitudinal measurements with HR-pQCT: evaluation of a 3D registration method to improve bone microarchitecture and strength measurement reproducibility. Bone. 2014 Jun;63:147-57. doi: 10.1016/j.bone.2014.03.001. Epub 2014 Mar 12. PMID 24614646
- [Background] Moller Dohn U, Boonen A, Hetland ML, Hansen MS, Knudsen LS, Hansen A, Madsen OR, Hasselquist M, Moller JM, Ostergaard M. Erosive progression is minimal, but erosion healing rare, in patients with rheumatoid arthritis treated with adalimumab. A 1 year investigator-initiated follow-up study using high-resolution computed tomography as the primary outcome measure. Ann Rheum Dis. 2009 Oct;68(10):1585-90. doi: 10.1136/ard.2008.097048. Epub 2008 Nov 19. PMID 19019887
- [Background] Finzel S, Rech J, Schmidt S, Engelke K, Englbrecht M, Stach C, Schett G. Repair of bone erosions in rheumatoid arthritis treated with tumour necrosis factor inhibitors is based on bone apposition at the base of the erosion. Ann Rheum Dis. 2011 Sep;70(9):1587-93. doi: 10.1136/ard.2010.148395. Epub 2011 May 27. PMID 21622765
- [Background] Dohn UM, Ostergaard M, Bird P, Boonen A, Johansen JS, Moller JM, Hansen MS. Tendency towards erosive regression on magnetic resonance imaging at 12 months in rheumatoid arthritis patients treated with rituximab. Ann Rheum Dis. 2009 Jun;68(6):1072-3. doi: 10.1136/ard.2008.098962. No abstract available. PMID 19435723
- [Background] Dohn UM, Ejbjerg B, Boonen A, Hetland ML, Hansen MS, Knudsen LS, Hansen A, Madsen OR, Hasselquist M, Moller JM, Ostergaard M. No overall progression and occasional repair of erosions despite persistent inflammation in adalimumab-treated rheumatoid arthritis patients: results from a longitudinal comparative MRI, ultrasonography, CT and radiography study. Ann Rheum Dis. 2011 Feb;70(2):252-8. doi: 10.1136/ard.2009.123729. Epub 2010 Oct 26. PMID 20980282
- [Background] Finzel S, Rech J, Schmidt S, Engelke K, Englbrecht M, Schett G. Interleukin-6 receptor blockade induces limited repair of bone erosions in rheumatoid arthritis: a micro CT study. Ann Rheum Dis. 2013 Mar;72(3):396-400. doi: 10.1136/annrheumdis-2011-201075. Epub 2012 May 14. PMID 22586162
- [Background] Garnero P, Thompson E, Woodworth T, Smolen JS. Rapid and sustained improvement in bone and cartilage turnover markers with the anti-interleukin-6 receptor inhibitor tocilizumab plus methotrexate in rheumatoid arthritis patients with an inadequate response to methotrexate: results from a substudy of the multicenter double-blind, placebo-controlled trial of tocilizumab in inadequate responders to methotrexate alone. Arthritis Rheum. 2010 Jan;62(1):33-43. doi: 10.1002/art.25053. PMID 20039425